CLINICAL TRIAL: NCT07215585
Title: A Phase III, Multicentre, Open-Label, Randomised Study Evaluating the Efficacy and Safety of R-mini-CHOP x2 Followed by AZD0486 Versus R-mini-CHOP x6 in Elderly or Unfit Participants With Newly Diagnosed Large B-cell Lymphoma (SOUNDTRACK-D2)
Brief Title: AZD0486 1L Therapy for Elderly or Unfit Participants With LBCL
Acronym: SOUNDTRACK-D2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D7402C00001; 2025-522029-37-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2025-10-07; First posted 2025-10-10 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Large B-cell Lymphoma
Keywords: Large B-cell Lymphoma; LBCL; AZD0486; CD3; CD19; TCE; B-cell malignancies; Soundtrack-D2

STUDY DESIGN:
Intervention Model Description: The study consists of 2 sequential parts: a safety run-in (SRI) followed by the phase III.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase III Arm A: R-mini-CHOP and AZD0486 (Experimental): 2 cycles of R-mini-CHOP followed sequentially by multiple cycles of AZD0486 at RP3D.
  Interventions: Drug: AZD0486; Drug: R-mini-CHOP
- Phase III Arm B: R-mini-CHOP (Active Comparator): 6 cycles of R-mini-CHOP per SoC regimen.
  Interventions: Drug: R-mini-CHOP
- Safety Run in: R-mini-CHOP and AZD0486 (Experimental): 2 cycles of R-mini-CHOP followed sequentially by multiple cycles of AZD0486 at RP2D.
  Interventions: Drug: AZD0486; Drug: R-mini-CHOP

INTERVENTIONS:
Drug: AZD0486 — Bispecific monoclonal IgG4 antibody
  Other Names: TNB-486
  Arms: Phase III Arm A: R-mini-CHOP and AZD0486; Safety Run in: R-mini-CHOP and AZD0486
Drug: R-mini-CHOP — Intravenous administration: Rituximab 375 mg/m2, Cyclophosphamide 400 mg/m2, Doxorubicin 25 mg/m2, Vincristine 1 mg, and Oral administration: Prednisone 40 mg/m2

SUMMARY:
The purpose of this study is to measure the efficacy and safety of R-mini-CHOP × 2 followed by AZD0486 compared with R-mini-CHOP × 6 in elderly or unfit participants newly diagnosed with LBCL.

ELIGIBILITY:
Inclusion criteria:

* Participants are either 80 years of age or older, OR 65 to 79 years of age or older and classified as unfit per sGA, and otherwise not considered candidates for full-dose R-CHOP per investigator assessment;
* Histologically confirmed diagnosis of previously untreated LBCL as per WHO-HEM5 (excluding plasmablastic lymphoma) and follicular large cell lymphoma;
* FDG-avid and measurable disease as per Lugano and Ann Arbor staging;
* Stage I bulky (7.5 cm and greater) to Stage IV;
* ECOG performance status 0 to 2;
* Adequate bone marrow, liver, renal and cardiac function.

The above is a summary, other inclusion criteria details may apply.

* As judged by the investigator, any evidence of diseases which make it undesirable for the participant to participate in the study, or that would jeopardise compliance with the protocol
* Diagnosis of post-transplant lymphoproliferative disease, plasmablastic lymphoma, Richter's transformation, prior history of or concurrent indolent lymphoma (including de novo transformed or composite lymphoma).
* History of CNS involvement by their B-NHL or history of clinically relevant CNS medical condition
* Known history of hemophagocytic lymphohistiocytosis/macrophage activation syndrome (HLH/MAS).
* Active or uncontrolled infection
* Major cardiac abnormalities
* Prior anti-lymphoma therapy except for corticosteroids for symptom control
* Requires chronic immunosuppressive therapy for active autoimmune/inflammatory condition, with some exceptions

The above is a summary, other exclusion criteria details may apply.

Ages: 65 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2030-07-09 (Estimated); Study Completion 2033-07-28 (Estimated)

PRIMARY OUTCOMES:
SRI - Safety evaluation of R-mini-CHOP × 2 followed by AZD0486: Number of participants with treatment-related adverse events. | Up to 1 year
  Incidence and severity of AEs, SAEs, AESIs, and events of clinical interest based on NCI CTCAE v5.0/ASTCT, vital signs, laboratory parameters.
SRI - Tolerability evaluation of R-mini-CHOP × 2 followed by AZD0486: Number of participants with treatment-related adverse events. | Up to 1 year
  AEs leading to study treatment discontinuation or dose modification based on NCI CTCAE v5.0/ASTCT, vital signs, laboratory parameters.
SRI - Determination of the recommended Phase III dose (RP3D) | Up to 1 year
  The RP3D will be the dose of AZD0486 selected for the Phase 3 part based on safety data compiled during the Safety Run-In part
Phase 3 - To demonstrate the superiority of R-mini-CHOP x2 followed by AZD0486 compared to R-mini-CHOP x6 regimen. | Up to 7 years
  Progression-free Surival (PFS), based on Lugano 2014 Response Criteria.

SECONDARY OUTCOMES:
Safety Run-In and Phase 3 - ORR | Up to 7 years
  ORR defined as the proportion of participants achieving either a PR or CR at timepoints defined in the study protocol, based on Lugano 2014 Response Criteria as determined by Investigator assessment.
Safety Run-In and Phase 3 - CR Rate | Up to 7 years
  CR rate is defined as the proportion of participants achieving a CR at timepoints defined in the study protocol, based on Lugano 2014 Response Criteria as determined by Investigator assessment.
Safety Run-In and Phase 3 - DoR | Up to 7 years
  DoR is defined as the time from the date of first documented response until the date of documented progression based on Lugano 2014 criteria as determined by Investigator assessment or death due to any cause.
Safety Run-In and Phase 3 - DoCR | Up to 7 years
  DoCR is defined as the time from the date of first documented CR until the date of documented progression or death due to any cause, as assessed by the Investigator.
Safety Run-In and Phase 3 - PFS | Up to 7 years
  PFS is defined as the time from date of the first dose to date of documented objective disease progression as per Lugano 2014 or death (by any cause in the absence of progression), as determined by Investigator assessment.
Safety Run In and Phase 3 - OS | Up to 7 years
  OS defined as the time from date of the first dose until death due to any cause.
Phase 3 - Time from randomisation to second progression or death (PFS2) | Up to 7 years
  PFS2 is defined as the time from randomisation to the earliest of the progression event (following the initial investigator-assessed progression), after first subsequent therapy, or death.
Phase 3 - Time to First Subsequent Therapy or Death (TFST) | Up to 7 Years
  TFST is defined as time from randomisation until the start date of first subsequent anti-lymphoma therapy after discontinuation of randomised treatment, or death due to any cause.
Phase 3 - Safety evaluation of R-mini-CHOP × 2 followed by AZD0486: Number of participants with treatment-related adverse events. | Up to 7 years
  Incidence and severity of AEs, SAEs, AESIs, and events of clinical interest based on NCI CTCAE v5.0/ASTCT, vital signs, laboratory parameters.
Phase 3 - Tolerability evaluation of R-mini-CHOP × 2 followed by AZD0486: Number of participants with treatment-related adverse events. | Up to 7 years
  AEs leading to study treatment discontinuation or dose modification based on NCI CTCAE v5.0/ASTCT, vital signs, laboratory parameters.
Safety Run-In and Phase 3 - Pharmacokinetics of AZD0486: serum concentration of study drug | Up to 7 years
  Maximum observed serum concentration of AZD0486.
Safety Run-In and Phase 3 - Pharmacokinetics of AZD0486: Maximum plasma concentration of the study drug (Cmax). | Up to 7 years
  Maximum observed plasma concentration of AZD0486.
Safety Run-In and Phase 3 - Pharmacokinetics of AZD0486: Concentration of study drug reached before next dose (Ctrough). | Up to 7 years
  Observed plasma concentration of AZD0486 right before next dose of AZD0486.
Safety Run-In and Phase 3 - To determine the immunogenicity of AZD0486 | Up to 7 years
  Summary of pre-existing and treatment induced ADAs for AZD0486 (positive or negative, titres) and the impact on PK, efficacy or safety.
Phase 3 - Safety evaluation of R-mini-CHOP × 2 followed by AZD0486 versus R-mini-CHOP × 6 | Up to 7 years
  Evaluation of key participant-reported side effects (pain, fatigue) and overall treatment tolerability, lymphoma-specific concerns, and HRQoL.
Phase 3 - Efficacy evaluation of R-mini-CHOP × 2 followed by AZD0486 versus R-mini-CHOP × 6 | Up to 7 years
  Evaluation of key participant-reported side effects (pain, fatigue) and overall treatment tolerability, lymphoma-specific concerns, and HRQoL.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dickinson,, MBBS BS DMSc, Principal Investigator — Peter MacCallum Cancer Center
Locations (38):
- Australia (2):
  - Research Site, Melbourne
  - Research Site, Nedlands
- Belgium (6):
  - Research Site, Antwerp
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Roeselare
  - Research Site, Yvoir
- Brazil (2):
  - Research Site, Porto Alegre
  - Research Site, São Paulo
- Canada (2):
  - Research Site, Calgary, Alberta
  - Research Site, Ottawa, Ontario
- China (7):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Nanchang
  - Research Site, Shandong
  - Research Site, Shanghai
- Hong Kong (3):
  - Research Site, Hong Kong
  - Research Site, Lai Chi Kok
  - Research Site, Shatin
- Japan (6):
  - Research Site, Bunkyō City
  - Research Site, Kōtoku
  - Research Site, Osaka
  - Research Site, Sunto-gun
  - Research Site, Yamagata
  - Research Site, Yokohama
- Poland (5):
  - Research Site, Kielce
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Wroclaw
- Research Site, Seoul, South Korea
- Turkey (Türkiye) (2):
  - Research Site, Ankara
  - Research Site, Antalya
- United Kingdom (2):
  - Research Site, London
  - Research Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home